CLINICAL TRIAL: NCT06196255
Title: Efficacy and Safety Study of Anti-FcRL5 CAR-T Cells in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: Safety and Efficacy of Anti-FcRL5 CAR-T Cell Therapy in Treating Relapsed and Refractory Multiple Myeloma (R/R MM)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, professor, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2023-KL216-01
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; FcRL5
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti FcRL5 CAR-T (Experimental): anti-FcRL5 autologous CAR T cells will be infused at a dose ranging from 1 - 2 x 10^6/kg CAR+ T cells after receiving lymphodepleting chemotherapy.
  Interventions: Drug: anti-FcRL5 CAR-T

INTERVENTIONS:
Drug: anti-FcRL5 CAR-T — anti-FcRL5 autologous CAR T cells will be infused at a dose ranging from 1 - 2 x 10^6/kg CAR+ T cells after receiving lymphodepleting chemotherapy.

SUMMARY:
This is an open label, single-arm, Phase 2 study to evaluate the efficacy and safety of Anti-FcRL5 CAR-T in subjects with relapsed and refractory multiple myeloma. A leukapheresis procedure will be performed to manufacture. Anti-FcRL5 chimeric antigen receptor (CAR) modified T cells. Prior to Anti-FcRL5 infusion subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide.

DETAILED DESCRIPTION:
This open label, single-arm, Phase 2 study aims to evaluate the efficacy and safety of Anti-FcRL5 CAR-T in subjects with relapsed and refractory multiple myeloma. A leukapheresis procedure will be performed to manufacture. Anti-FcRL5 chimeric antigen receptor (CAR) modified T cells. Prior to Anti-FcRL5 infusion subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide. After infusion, the investigators will observe the characteristics of dose limited toxicity (DLT), and determine the maximum tolerable agent MTD and rp2d were confirmed. To provide basis for the dosage and treatment plan of cell products in follow-up clinical trials.

ELIGIBILITY:
Inclusion Criteria:

The set subject inclusion criteria include multiple documents of multiple myeloma, no effective treatment options (e. g. autologous or allogeneic stem cell transplantation) and limited outcome (<2 years) with existing therapies, as follows:

1. Age is 18~70 years old;
2. Expected survival period of>12 weeks;
3. Multiple myeloma was diagnosed by physical examination, pathological examination, laboratory examination and imaging;
4. Patients with refractory multiple myeloma;
5. Patients with multiple myeloma recurrence;
6. ALT and AST <3 times normal; bilirubin <2.0mg / dl;
7. Quality of survival score (KPS)> 50%;
8. The patient has no serious heart, liver, kidney and other diseases;
9. Recurrence or no disease remission after hematopoietic stem cell transplantation or cellular immunotherapy;
10. Is not suitable for stem cell transplantation conditions or to abandon transplantation due to conditional restrictions;
11. Blood can be obtained intravenously, without other contraindications to leukapheresis;
12. Understand and voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding, or who have a pregnancy plan within six months;
2. Infectious diseases (such as HIV, active tuberculosis, etc.);
3. Active hepatitis B or hepatitis C infection;
4. Feasibility assessment screening demonstrated <10% transfection of targeted lymphocytes or underamplification under CD3 / CD28 costimulation (<5-fold);
5. Abnormal vital signs, and unable to cooperate with the examination;
6. Have mental or mental illness who cannot cooperate with the treatment and efficacy evaluation;
7. Highly allergic constitution or have a history of severe allergies, especially allergic to IL-2;
8. Subjects with a systemic infection or a severe local infection requiring anti-infective treatment;
9. Subjects with severe autoimmune disease;
10. The doctor believes there were other reasons for inclusion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-12-25 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Baseline up to 28 days after CAR-T cells infusion
  Adverse events assessed according to NCI-CTCAE v5.0

SECONDARY OUTCOMES:
overall response rate (ORR) | Month 6, 12, 18 and 24
  Assessment of ORR at Month 6, 12, 18 and 24
complete response (CR) | Month 6, 12, 18 and 24
  Assessment of CR at Month 6, 12, 18 and 24
Overall survival (OS) | Month 6, 12, 18 and 24
  Assessment of OS at Month 6, 12, 18 and 24
Event-free survival (EFS) | Month 6, 12, 18 and 24
  Assessment of EFS at Month 6, 12, 18 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Kailin Xu, MD.,PD., Study Chair — The Affiliated Hospital oh Xuzhou Medical University
Locations (1):
- The affiliated hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No